CLINICAL TRIAL: NCT01434056
Title: Prediction of Mortality in Patients Waiting for Liver Transplantation Through Brain Magnetic Resonance Imaging
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Principal Investigator, Ellison Fernando Cardoso, MD, PhD, Hospital Israelita Albert Einstein
Other Study IDs: 1341-11; CEP1572 (Other: Ethical Committee Research)
Record Dates: First submitted 2011-09-13; First posted 2011-09-14 (Estimated); Last update posted 2011-09-14 (Estimated); Status verified 2011-09

CONDITIONS: End Stage Liver Disease; Hepatic Encephalopathy
Keywords: Liver disease; Hepatic encephalopathy; MELD; Liver transplantation
MeSH Terms: conditions — End Stage Liver Disease; Hepatic Encephalopathy; Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Liver transplantation waiting list: Patients waiting for liver transplantation with chronic end staged liver disease

SUMMARY:
The purpose of this study is to determine whether hepatic encephalopathy, measured through magnetic resonance imaging, electroencephalogram and neuropsychological evaluation adds prognostic information to patients who are waiting for liver transplantation. If this model improves mortality prediction this might be used in the future for organ allocation.

DETAILED DESCRIPTION:
The only current definitive treatment for end-stage liver disease is transplantation. Due to the scarcity of organs available, the correct prioritization of patients for liver transplantation has a crucial importance. Nowadays, patients are ranked according to severity of liver disease, measured by the MELD score. This index is only derived from objective measures (serum concentration of bilirubin, creatinine and INR). Hepatic encephalopathy (HE) is a serious and progressive disorder in patients with end-stage liver disease. The severity of HE has prognostic implications in those waiting for liver transplantation. However, the prognosis of HE is independent and not correlated to the MELD score. Hepatic encephalopathy triggers multiple changes in brain magnetic resonance imaging (MRI) providing an objective way to evaluate it. Also electroencephalogram and neuropsychological evaluation might increase mortality prediction.

Adding the information provided by MRI, electroencephalogram and neuropsychological evaluation to the MELD score model might increase the prediction of mortality. Increase mortality's prediction has a fundamental importance because in organ allocation.

We will evaluate the predictive value of these variables in predicting mortality of those patients waiting for liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman over 18 years old
* Listed in liver transplantation waiting line
* Patient able and willing to participate in the evaluations of this study

Exclusion Criteria:

* Acute liver failure
* Serious structural brain anomalies
* Condition or situation in which, in the opinion of the investigator, put the patient at significant risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients waiting for liver transplantation with chronic end stage liver disease.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2011-11; Primary Completion 2014-11 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Mortality | Three months

CONTACTS AND LOCATIONS:
Overall Officials: Edson Amaro Junior, MD,PhD, Study Chair — Hospital Israelita Albert Einstein
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Habib S, Berk B, Chang CC, Demetris AJ, Fontes P, Dvorchik I, Eghtesad B, Marcos A, Shakil AO. MELD and prediction of post-liver transplantation survival. Liver Transpl. 2006 Mar;12(3):440-7. doi: 10.1002/lt.20721. PMID 16498643